CLINICAL TRIAL: NCT00863707
Title: A Phase 4, Multicenter, Double-Blind, Randomized, Placebo-controlled Study of the Safety and Tolerance of Regadenoson in Subjects With Renal Impairment
Brief Title: A Study of the Safety and Tolerance of Regadenoson in Subjects With Renal Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3606-CL-3010
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Results first posted 2011-01-31 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Kidney Diseases; Coronary Artery Disease
Keywords: regadenoson; chronic kidney disease stage III; chronic kidney disease stage IV; renal impairment; coronary artery disease
MeSH Terms: conditions — Kidney Diseases; Coronary Artery Disease; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — regadenoson

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matching intravenous (IV) bolus injection
  Interventions: Drug: Placebo
- Regadenoson (Experimental): 0.4 mg/5 mL intravenous bolus injection
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — IV
  Other Names: CVT-3146; Lexiscan
  Arms: Regadenoson
Drug: Placebo — IV
  Arms: Placebo

SUMMARY:
This study is intended to assess the safety and tolerance of regadenoson in subjects with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Stage III or Stage IV renal impairment based on the National Kidney Foundation (NKF) Kidney Disease Outcomes Quality Initiative (K/DOQI) glomerular filtration rate (GFR) classification
* Subject has a diagnosis of Coronary Artery Disease (CAD) or risk factors for CAD as determined by a current medical diagnosis of at least 2 of the following conditions: Type 2 diabetes, hypertension, hypercholesterolemia, current or history of cigarette smoking (minimum 10 pack-years exposure) or obesity (Body Mass Index (BMI) > 30)
* Subject must abstain from smoking 3 hours prior and 8 hours post study drug administration
* Subject must abstain from any intake of foods and beverages containing a methylated xanthine derivative (i.e. caffeine, theobromine, or methylxanthine) within 12 hours prior to study drug administration through the Follow-Up visit, as these foods may reduce the effects of regadenoson derivative (i.e. caffeine, theobromine, or methylxanthine) within 12 hours prior to study drug administration through the Follow-Up visit, as these foods may reduce the effects of regadenoson

Exclusion Criteria:

* Subject has a history of an additional clinically significant illness, medical condition, or laboratory abnormality within 2 weeks prior to Screening
* Female subject who is pregnant, lactating or of childbearing potential who refuses to use a medically acceptable form of contraception until the Follow-Up visit is complete

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development
Locations (39):
- United States (39):
  - Anniston, Alabama
  - Little Rock, Arkansas
  - Bell Gardens, California
  - Fullerton, California
  - Garden Grove, California
  - Los Angeles, California
  - Mission Viejo, California
  - Oakland, California
  - Roseville, California
  - Santa Ana, California
  - Newark, Delaware
  - Wilmington, Delaware
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Orlando, Florida
  - Trinity, Florida
  - Winter Park, Florida
  - Ellijay, Georgia
  - Chicago, Illinois
  - Auburn, Maine
  - Detroit, Michigan
  - Flint, Michigan
  - Minneapolis, Minnesota
  - Ridgewood, New Jersey
  - Somerset, New Jersey
  - New York, New York
  - Springfield Gardens, New York
  - Springfield, Ohio
  - Oklahoma City, Oklahoma
  - Bend, Oregon
  - Duncansville, Pennsylvania
  - Indiana, Pennsylvania
  - Tyrone, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Spartanburg, South Carolina
  - Knoxville, Tennessee
  - Houston, Texas
  - Sugar Grove, Texas

REFERENCES:
- [Background] Ananthasubramaniam K, Weiss R, McNutt B, Klauke B, Feaheny K, Bukofzer S. A randomized, double-blind, placebo-controlled study of the safety and tolerance of regadenoson in subjects with stage 3 or 4 chronic kidney disease. J Nucl Cardiol. 2012 Apr;19(2):319-29. doi: 10.1007/s12350-011-9508-3. Epub 2012 Jan 19. PMID 22259009
- See also: Link to Prescribing Information — http://www.astellas.us/docs/lexiscan.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Regadenoson
Started | 174 | 337
Completed | 170 (Completed Population is equal to Safety Analysis Set (SAF)) | 334 (Completed Population is equal to Safety Analysis Set (SAF))
Not Completed | 4 | 3
Not completed — Randomized, but drug not received | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Regadenoson | Total
Number analyzed (Participants) | 170 | 334 | 504
Age Continuous [Mean (Standard Deviation); unit: years] | 66.1 (10.91) | 66.4 (11.25) | 66.3 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 150 | 228
  Male | 92 | 184 | 276
Race/Ethnicity, Customized [Number; unit: participants]
  White | 115 | 254 | 369
  Black or African American | 47 | 68 | 115
  Asian | 6 | 10 | 16
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian - Other Pacific Islander | 1 | 0 | 1
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subject With Serious Treatment Emergent Adverse Events (TEAE)
Description: The data represents the numbers of subjects reporting Serious TEAEs.
  TEAEs were defined as Adverse Events (AEs) starting or worsening after administration of the test drug.
Time Frame: 24 hours post dose
Population: The number of participants analyzed per arm represents Safety Analysis Set (SAF); all randomized subjects who received any amount of study drug.
Measure: Number; unit: Subjects
Arm/Group | Placebo | Regadenoson
Number analyzed (Participants) | 170 | 334
Subjects | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event collection began immediately following study drug administration through the follow-up visit. All Serious Adverse Events (SAEs) occurring until 30 days after dosing were reported.
Description: TEAEs were defined as AEs starting or worsening after starting administration of the test drug.
  Within a system organ class subjects may have reported more than one type of Adverse Event.
Arm/Group | Placebo | Regadenoson
Serious Adverse Events (participants affected / at risk) | 1/170 | 0/334
Other Adverse Events (participants affected / at risk) | 20/170 | 184/334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=170) | Regadenoson (N=334)
Death (Cardiac disorders) | 1 | 0 — SAE Investigator Reported Term "Pulmonary Cardiac Arrest" coded to "Death" was reported after the follow-up visit.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=170) | Regadenoson (N=334)
Headache (Nervous system disorders) | 12 | 83
Dizziness (Nervous system disorders) | 1 | 32
Dysgeusia (Nervous system disorders) | 6 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 64
Nausea (Gastrointestinal disorders) | 2 | 49
Chest discomfort (General disorders) | 1 | 49
Flushing (Vascular disorders) | 3 | 40

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.